CLINICAL TRIAL: NCT06265753
Title: Effects of Gastrocinemius Function Massage on Lower Extemity Spasticity, Spatio- Temporal Gait Variables and Fall Risk ın Patients With Stroke
Brief Title: Gastrocinemius Function Massage on Lower Extemity Spasticity
Acronym: Spasticity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Emre BASKAN, Assoc. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gastrocimemius spasticity; E-60116787-020-474196 (Registry Identifier: Pamukkale University Ethics Comitee)
Record Dates: First submitted 2024-01-24; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Stroke Ischemic
Keywords: Spacticity, Gastrocinemius function massage, stroke, gait
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: In the study, 2 different groups (experimental and control) will be formed by using randomisation method. In addition to 45 minutes of classical physiotherapy exercises, 10 minutes of gastrocinemius function massage will be applied to the experimental group, while 10 minutes of sham massage and 45 minutes of classical physiotherapy exercises will be applied to the control group. The application will continue 2 days a week for 6 weeks. Spasticity, gait parameters and fall risks of the participants will be evaluated before and after the treatment with the help of various tests.
  Translated with www.DeepL.com/Translator (free version)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Who received 10 minutes gastrocinemius function massage and 45 minutes classic physiotherapy exercise
  Interventions: Other: Gastrocinemius Function Massage
- Control group (Sham Comparator): Who received 10 sham applicaiton massage and 45 minutes classic physiotherapy exercise
  Interventions: Other: Sham application

INTERVENTIONS:
Other: Gastrocinemius Function Massage — The purpose of gastrocnemius massage is to alleviate muscle stiffness in the gastrocnemius muscle and enhance mobility in the foot and ankle of the individuals involved. During the GFM application, the patient assumes a prone posture on a suitable treatment bed. The therapist positions themselves behind the patient's side and secures the patient's foot between their hip and ilium.The therapist firmly holds the gastrocnemius muscle using both hands and applies pressure to the ankle, causing it to move in the direction of dorsiflexion. Simultaneously, the therapist applies mobilisation in the cranial direction, following the same path as the gastrocnemius muscle fibres, using both hands. Afterwards, the therapist gently pulls the arm and trunk backwards until the foot and gastrocnemius muscle become relaxed. The application is sustained in a rhythmic manner . We will apply this massage aproximately 10 min to experimental group.
  Arms: Experimental Group
Other: Sham application — The sham application was conducted when the patient was lying face down, with the hands placed on the gastrocnemius muscle without any movement. We will apply this application aproximately 10 min to experimental group.
  Arms: Control group

SUMMARY:
This study aimed to investigate gastrocinemius function massage on physical parameters of stroke patients.

DETAILED DESCRIPTION:
Gastrocinemius function massage is known to relieve pain and increase range of motion. However, its effects on spasticity and physical performance in stroke patients are not fully understood. In this study, we aimed to investigate the effects of gastrocinemius function massage.

ELIGIBILITY:
Inclusion Criteria:

* having experienced a stroke at least 6 months prior,
* being able to stand independently for at least 1 minute,
* scoring at least 23 on the Standardised Mini-Mental State Examination (SMMSE), indicating no significant cognitive impairment , and
* having lower extremity spasticity rated between 1-3 on the modified Asworth scale
* at least 18 years of age.

Exclusion Criteria:

* comorbidities such as neurological, orthopaedic, metabolic, and rheumatological diseases that could potentially impact soft tissues.
* patients who had received spasticity or other treatments that could affect soft tissues within the past 3 months,
* those with lower extremity injuries, and those with a diagnosis of cancer or who were pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Spasticity | aproximately 10 miutes
  Modified Aswort Scale is used to asses spasticity level of participants,The Muscle Assessment Scale (MAS) is a method utilised to assess the degree of resistance experienced during passive range of motion exercises. This evaluation does not necessitate any specialised equipment and can be conducted swiftly (Bohannon and Smith, 1987). The assessment of the efficacy of pharmacological and rehabilitative therapies in the treatment and management of spasticity in stroke patients is commonly employed (Ansasri et al., 2008). The scale is denoted by the subsequent numerical values (Ansasri et all., 2008). 0: Absence of increase in muscular tone 1: There is a little rise in muscle tension, accompanied by a mild resistance or moderate challenge at the furthest point of movement when flexing or extending the affected body part(s). 1+: A slight augmentation in muscular tension is succeeded by negligible opposition throughout the remaining (less than 50%) of the motion range.
Gait parameters and fall risk | aproximately 5 miutes
  Spatial Temporal Gait Analysis, also known as Legsystm, is a method used to analyse the movement patterns and timing of an individual's gait. The walking variables of the subjects were assessed using a wearable walking analysis device known as Legsystm. The user's text is empty. The data gathered by two sensors affixed to the supramaleo region using Velcro is transmitted and processed to the connected computer using Bluetooth. Legsystm possesses the capacity to perform diverse measurements of spatio-temporal data obtained from people. During the Legsystm analysis, participants were instructed to perform the Time up and go test. The Timed Up and Go (TUG) test will be utilised to evaluate the spatio-temporal parameters and ascertain the likelihood of falling in stroke patients. During the TUG (Timed Up and Go) test, the patient is initially positioned in an appropriate chair.

CONTACTS AND LOCATIONS:
Locations (1):
- University Address, Denizli, Muş Alparslan University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dengiz A, Sekeroz S, Baskan E, Kara G. Effects of gastrocnemius functional massage on lower extemity spasticity, spatio- temporal gait variables and fall risk in patients with stroke: A randomized controlled trial. PLoS One. 2025 Sep 24;20(9):e0332308. doi: 10.1371/journal.pone.0332308. eCollection 2025. PMID 40991570